CLINICAL TRIAL: NCT01260558
Title: Pilop Trial of OCT-determined Coverage of Permanent or Polymer-free Sirolimus Eluting Stent at Long Term
Brief Title: Test of Long-Term Safety and Efficacy of Sirolimus-Permanent-Polymer Eluting Stent (Cypher)- and Sirolimus-Polymer-free Eluting Stents (PPS/PFS) Assessed by Optical Coherence Tomography
Acronym: PPS/PFS-OCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S03310
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Sirolimus-Permanent-Polymer Eluting Stent
  Interventions: Device: Sirolimus-Permanent-Polymer Eluting Stent
- Arm 2 (Active Comparator): Sirolimus-Polymer-free Eluting Stent
  Interventions: Device: Sirolimus-Polymer-free Eluting Stent

INTERVENTIONS:
Device: Sirolimus-Permanent-Polymer Eluting Stent — due randomization sirolimus-permanent-polymer eluting stent was implanted
  Other Names: Cypher®
  Arms: Arm 1
Device: Sirolimus-Polymer-free Eluting Stent — due randomization sirolimus-polymer-free eluting stent was implanted
  Other Names: ISAR Rapa G1
  Arms: Arm 2

SUMMARY:
The objective of this pilot study is to compare the PFS-eluting stent (ISAR Rapa G1) with the PPS-eluting stent (Cypher®) regarding uncovered stent strut segments at 5 years.

DETAILED DESCRIPTION:
The mid-term efficacy of drug-eluting stents has been well-established, but there is an ongoing debate on the potential of an increased incidence of late stent thrombosis, particularly after discontinuation of thienopyridine therapy, as well as of delayed onset of restenosis or catch-up phenomenon with permanent polymer-based DES. The extent of strut coverage with reduction of exposed thrombogenic material has been shown to be associated with the inflammatory reaction grade and with the incidence of stent thrombosis. The optical coherence tomography (OCT) is an intravascular imaging modality based on light. The principle is similar to intravascular ultrasound, but due to the much shorter wave length of light, it offers a much better resolution up to 10µm, enabling the exact determination of strut coverage, neointimal thickness, vessel size, presence of dissections, and even the presence of inflammation.

Patients who received a polymer-free or a permanent-polymer sirolimus-eluting stent about 5 years ago without in-segment intervention since, will be evaluated by OCT regarding the healing pattern and the late lumen loss of the stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with with previous implantation of polymer-free or permanent-polymer sirolimus-eluting stents 5 years ago due to ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% stenosis located in native coronary vessels.
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study and assessment by OCT.
* In women with childbearing potential a negative pregnancy test is mandatory.

Exclusion Criteria:

* Intervention in the segment of the study stent after the index procedure
* Target lesion located in the left main trunk.
* In-stent restenosis with difficulty to pass the OCT device
* Acute myocardial infarction
* Known allergy to the study medications: Sirolimus, rapamycin, probucol or stainless steel.
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Degree of stent strut coverage after 5 years assessed by OCT for each visible strut segment | 5 years

SECONDARY OUTCOMES:
Percentage of malapposed strut assessed by OCT | 5 years
Percentage of uncovered malapposed struts assessed by OCT | 5 years
Morphologic differences of neointima between stents | 5 years
Late lumen loss at 5 years assessed by OCT | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Tiroch, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich, Bavaria
  - Klinikum rechts der Isar, Munich, Bavaria